CLINICAL TRIAL: NCT01947036
Title: T and B Cell Responses Across Autoimmune Diseases
Brief Title: T and B Cell Responses in Autoimmune Diseases
Acronym: SRA01
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT SRA01
Record Dates: First submitted 2013-09-16; First posted 2013-09-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes Mellitus; Multiple Sclerosis; Arthritis, Rheumatoid; Crohn's Disease; Psoriasis
Keywords: autoimmune disease; immune-mediated disease; T and B cells immunophenotype; IL23 signaling; genetic risk variants
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Multiple Sclerosis; Arthritis, Rheumatoid; Crohn Disease; Psoriasis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Healthy Subjects: Healthy adult controls (no auto-immune disease)
- Subjects with Crohn's Disease: Diagnosed with or suspected of having Crohn's disease (CD)
- Subjects with Rheumatoid Arthritis: Diagnosed with or suspected of having rheumatoid arthritis (RA)
- Subjects with Type 1 diabetes: Diagnosed with or suspected of having type 1 diabetes mellitus (T1D, T1DM)
- Subjects with Multiple Sclerosis (MS): Diagnosed with or suspected of having MS
- Subjects with Psoriasis: Diagnosed with or suspected of having psoriasis (Ps)

SUMMARY:
The study aims to establish whether defects in immune cell function are shared across multiple autoimmune diseases and whether those problems match to similar genes in the cells.

DETAILED DESCRIPTION:
This is a non-randomized, multi-center clinical research study. Subjects who are healthy or have a confirmed or suspected diagnosis of type 1diabetes, multiple sclerosis, psoriasis, Crohn's disease, or rheumatoid arthritis will be asked to donate a blood sample. No follow-ups are planned.

Investigators will:

* evaluate immune cells from subjects enrolled in this study and match the differences to types of immune cells known to cause autoimmune diseases
* investigate a particular disease pathway: the IL23R signaling cascade.

ELIGIBILITY:
Inclusion Criteria:

-Subject or subject's parent or legal guardian has provided written informed consent

-For healthy donors: Healthy individuals between 18 and 60 years of age, inclusive

* For all subjects with an autoimmune disease:

  1. Adults between 18 and 60 years, inclusive, diagnosed with or suspected of having one of the following five diseases: adult forms of rheumatoid arthritis (RA), type 1 diabetes (T1D, T1DM), multiple sclerosis (MS), Crohn's disease (CD), Psoriasis (Ps)
  2. Or Children from 8 years up to 18 years inclusive, diagnosed with or suspected of having type 1 diabetes (TID) or Crohn's disease (CD)
  3. Treatment naïve except for prednisone (or equivalent corticosteroid) <\=10mg/day

     4. For subjects diagnosed with type 1 diabetes:

  <!-- -->

  1. Clinical diagnosis or suspected diagnosis of T1D
  2. Positive per standard clinical titer levels for anti-insulin antibodies if within 10 days of diagnosis (new-onset T1D); and otherwise one of the following antibodies-anti-GAD65, anti-ICA512/IA2 or anti-ZnT8
  3. Minimum body weight 17kg (≥37.5 pounds)
  4. Disease duration within 1 year

     5. For subjects diagnosed with multiple sclerosis:

  a. EDSS (Expanded Disability Status Scale) 0-5 b. Diagnosis or suspected diagnosis of MS as per Dr. Polman et al. Annals of Neurology 2010 c. Disease duration within 1 year

  6. For subjects diagnosed with rheumatoid arthritis (RA):

  a. Diagnosis or suspected diagnosis of RA (2010 ACR criteria) b. Anti-CCP antibody positive c. Disease duration within 1 year

  7. For subjects diagnosed with Crohn's disease:

  a. Clinical diagnosis or suspected diagnosis of Crohn's confirmed by endoscopy b. Disease duration within 1 year c. Minimum body weight 17 kg (≥37.5 pounds)

  8. For subjects diagnosed with psoriasis:
  1. Psoriasis diagnosis by a dermatologist
  2. Disease duration within 1 year
  3. At least two psoriatic plaques or a single plaque occupying at least 1% of total body surface outside scalp

     Exclusion Criteria:

     1. For healthy donors:

  a. Individuals who are unable or unwilling to donate blood samples b. Individuals with self-reported chronic metabolic diseases such as type 2 diabetes, impaired glucose tolerance or morbid obesity c. Individuals with self-reported acute infection (respiratory or others) or chronic infection (such as HIV,hepatitis B or -C) d. Individuals with self-reported immune-mediated diseases such as multiple sclerosis, type 1 diabetes, primary immunodeficiency e. Individuals with self-reported current or prior history of malignancy f. Individuals who are currently pregnant (self-report) g. Corticosteroid therapy equivalent to >/= 10 mg/day of prednisone within the last 4 weeks h. Immunosuppressive therapy at any time prior to enrollment (such as Cyclophosphamide, Mitoxantrone, Imuran, Cellcept, Methotrexate, Rituximab, Alemtuzumab)

  2. For all subjects with an autoimmune disease:

  a. Pregnant patients b. Pediatric patients unable to donate at least 51 mL of blood per NIH guidelines (no more than 5 mL/kg in a single day and no more than 9.5 mL/kg over any 8 week period) c. Patients with current substance abuse or alcoholism (self-report) d. Patients diagnosed with more than one autoimmune and/or inflammatory disease, exception - asthma is permissible e. Corticosteroid therapy equivalent to > 10 mg/day of prednisone within the last 4 weeks f. Immunomodulatory therapies within the last 12 months (such as Interferon, Glatiramer Acetate, Natalizumab, Fingolimod) g. Immunosuppressive medication at any time prior to enrollment (such as Cyclophosphamide, Mitoxantrone, Imuran, Cellcept, Methotrexate, Rituximab, Alemtuzumab) h. Any prior or current Anti-tumor necrosis factor (anti-TNF) treatments i. Any prior or current use of experimental drugs tested in Phase I, II, or III clinical trials

  3. Diagnosis of ulcerative colitis or indeterminate colitis

  4. Pustular psoriasis, isolated palmoplantar psoriasis, isolated inverse psoriasis and isolated sebopsoriasis.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who are healthy or have a confirmed or suspected diagnosis of type 1 diabetes (T1D, T1DM), multiple sclerosis (MS), psoriasis (Ps), Crohn's disease (CD), or rheumatoid arthritis (RA) will be invited to donate a blood sample. No follow-ups are planned.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Identify shared defects in T and B cell function by disease classification | One-time blood draw
  The study aims to establish whether defects in T and B cell function are shared across multiple immune-mediated diseases and whether these are driven by shared genetic risk variants.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cotsapas, PhD, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Feinstein Institute for Medical Research, Manhasset, New York
  - University of Rochester, Rochester, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Baylor Institute of Immunology Research - Clinical Rheumatology, Dallas, Texas

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/